CLINICAL TRIAL: NCT02103751
Title: A Multi-center Study to Determine the Levels of Biomarkers of Potential Harm and Biomarkers of Exposure to Cigarette Smoke in Asian Adult Smokers and Non-smokers
Brief Title: Determination of Biomarkers of Exposure and Biomarkers of Potential Harm in Asian Adult Cigarette Smokers
Status: Completed | Type: Observational
Sponsor: Philip Morris Products S.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: CS06-01
Record Dates: First submitted 2014-03-20; First posted 2014-04-04 (Estimated); Last update posted 2019-11-07 (Actual); Status verified 2019-11

CONDITIONS: Smoking; Healthy
Keywords: biomarkers; HPHCs; CVD; smoking; Smokers; non-smokers
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to determine biomarkers of exposure to Harmful and Potentially Harmful Constituents (HPHCs) in Cigarette Smoke and cardiovascular-related biomarkers in smokers and non smokers.

DETAILED DESCRIPTION:
Since Japanese mortality associated with cardiovascular disease (CVD) is lower than that in the USA although Japan is one of the top four tobacco consuming countries, this study aims to determine biomarkers of both level of exposure and CVD-related biological effects in Japanese smokers compared to non-smokers.

Biomarkers of Exposure (BoExp) include 2-naphthylamine (2-NA), 4-aminobiphenyl (4-ABP), 4-(methylnitrosaminoi)-1-(3-pyridil)-1-butanone (NNK), carbon monoxide (CO), nicotine, pyrene and 0-toluidine (o-TOL). CVD-related biomarkers include white blood cell (WBC) count, high sensitivity C-reactive protein (hs-CRP) and homocysteine in plasma; complemented with urinary 8-epi-prostaglandin F2α (8-epi-PGF2α), plasma malondialdehyde (MDA), urinary 11-DTXB2, plasma fibrinogen, high-density lipoprotein-cholesterol, triglycerides, sICAM-1, sVCAM-1 and von Willebrand Factor.

ELIGIBILITY:
Inclusion Criteria:

* Smokers have smoked commercially available conventional cigarettes (CC)
* With a minimum consumption of 10 CC per day for the last 5 years

Exclusion Criteria:

* Any prior medical condition or chronic disease
* Recent infection
* History of cancer
* Use of concomitant medication
* History of alcohol abuse
* Pregnant women

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy male and female Japanese smokers and non smokers, 30 years of age or older.
Sampling Method: Probability Sample
Enrollment: 1069 (Actual)
Dates: Start 2007-07; Primary Completion 2007-12 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
The level of biomarkers of Exposure (BoExp) to HPHCs - present in cigarette smoke - in Asian smokers compared to non smokers | At Visit 2 (up to14 days after Visit 1)
  To measure the level of smoking, at baseline the Fagerstrom nicotine dependence test and urinary cotinine are measured. For measurement of biomarkers of exposure, blood and 24 hour urine sampling are performed at V2.
The level of CVD-related biomarkers in Asian smokers compared to non smokers | At Visit 2 (up to14 days after Visit 1)

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Tomoko Hasunuma, MD, Principal Investigator — Kitasato University, Tokyo, Japan
Locations (1):
- Bio-Iatric Centre, Research Institute for Clinical Pharmacology, Kitasato University, Tokyo, Japan

REFERENCES:
- [Result] Ludicke F, Magnette J, Baker G, Weitkunat R. A Japanese cross-sectional multicentre study of biomarkers associated with cardiovascular disease in smokers and non-smokers. Biomarkers. 2015;20(6-7):411-21. doi: 10.3109/1354750X.2015.1096303. PMID 26616146